CLINICAL TRIAL: NCT01528631
Title: Randomized Controlled Double-blind Nutritional Intervention Trial to Evaluate the Effects of D-fagomine on Glycaemic Response to Sucrose in Men
Brief Title: The Effects of D-Fagomine on Glycaemic Response to Sucrose in Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioglane (Industry)
Collaborators: University Rovira i Virgili (Other); Technological Centre of Nutrition and Health (Other); National Research Council, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1AP029010911
Record Dates: First submitted 2012-02-03; First posted 2012-02-08 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Glycaemic Response; Insulinemic Response
MeSH Terms: interventions — fagomine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Product (Placebo Comparator): 200 ml water with 50g of sucrose
  Interventions: Other: D-Fagomine
- Product 1 (Active Comparator): 200 ml water with 50g of sucrose and supplemented with 30 mg of D-Fagomine
  Interventions: Other: D-Fagomine

INTERVENTIONS:
Other: D-Fagomine — 30 mg (initial dose), with 50 grams of sucrose in 200 ml of water.
  Arms: Product 1
Other: D-Fagomine — 0 mg (control) blended with 50 grams of sucrose in 200 ml of water.
  Arms: Control Product

SUMMARY:
The aim of this study is to evaluate the effect of D-fagomine on glycaemic response to sucrose in men.

DETAILED DESCRIPTION:
To determine and compare glycaemic response to sucrose of D-Fagomine and control in the timeframe of 180 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Males between the ages of 20 and 70 willing and able to provide written informed consent.

Exclusion Criteria:

1. LDL cholesterol levels higher than 189 mg/dl
2. Triglycerides higher than 350 mg/dl (the threshold level to determine c-LDL using the Friedewald formula)
3. Physical examinations and routine biochemical analysis shall be conducted to rule out pathologies.
4. Consumption of supplements or acetylsalicylic acid
5. Chronic alcoholism
6. Body mass index (BMI) greater than 30 kg/m2
7. Previous antihypertensive treatment at the start of the trial that has not finished at least 2 months before beginning the study
8. Diabetes mellitus (if the fasting blood glucose is higher than 126 mg/dl, the test should be repeated and confirmed)
9. Kidney disease (serum creatine levels above 1,4 mg/dl for women and above 1,5 mg/dl for men)
10. Acute infectious diseases, malignant tumors, severe liver failure, respiratory failure associated with chronic or endocrine diseases
11. Other conditions such as special dietary needs
12. To be participating or having participated in a clinical trial within the last 3 months
13. Inability to continue the study
14. History of gastrointestinal disease which may alter the absorption of nutrients
15. Depressive disorder or thoughts of self-injury

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-02; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Glycaemic response to sucrose | 0-180 minutes

SECONDARY OUTCOMES:
Insulin in venous plasma | 0-180 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Solà, PhD MD, Principal Investigator — University Rovira i Virgili
Locations (1):
- Hospital Universitari Sant Joan, Universitat Rovira i Virgili, Reus, Tarragona, Spain

REFERENCES:
- [Background] Gomez L, Molinar-Toribio E, Calvo-Torras MA, Adelantado C, Juan ME, Planas JM, Canas X, Lozano C, Pumarola S, Clapes P, Torres JL. D-Fagomine lowers postprandial blood glucose and modulates bacterial adhesion. Br J Nutr. 2012 Jun;107(12):1739-46. doi: 10.1017/S0007114511005009. Epub 2011 Oct 3. PMID 22017795
- See also: BIOGLANE SLNE — http://www.bioglane.com
- See also: D-Fagomine — http://www.fagomine.com
- See also: CTNS - Technology Centre of Nutrition and Health — http://www.ctns.cat
- See also: URV - Rovira i Virgili University — http://www.urv.cat